CLINICAL TRIAL: NCT02871492
Title: A Randomized, Double-blind, Multi-center, Three Arm (Pritelivir, Placebo and Zovirax®) Parallel Group, Comparative Trial to Assess the Efficacy and Safety of Pritelivir 5% w/w Ointment for the Treatment of Recurrent Herpes Labialis in Adults - LipP1
Brief Title: Trial on Efficacy and Safety of Pritelivir Ointment for Treatment of Labial Herpes
Acronym: LipP1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AiCuris Anti-infective Cures AG (Industry)
Collaborators: Novella Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIC316-02-II-01
Record Dates: First submitted 2016-08-05; First posted 2016-08-18 (Estimated); Results first posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Herpes Labialis
Keywords: HSV, pritelivir, herpes, herpes labialis, topical,
MeSH Terms: conditions — Herpes Labialis; Herpes Simplex | interventions — pritelivir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pritelivir 5% w/w ointment (Experimental): Topical treatment (20 applications), 5 times daily for 4 days
  Interventions: Drug: Pritelivir 5% w/w ointment
- Pritelivir ointment matching placebo (Placebo Comparator): Topical treatment (20 applications), 5 times daily for 4 days
  Interventions: Drug: Pritelivir ointment matching placebo
- Zovirax® cream (Active Comparator): Topical treatment (20 applications), 5 times daily for 4 days
  Interventions: Drug: Zovirax® cream

INTERVENTIONS:
Drug: Pritelivir 5% w/w ointment
  Arms: Pritelivir 5% w/w ointment
Drug: Pritelivir ointment matching placebo
  Arms: Pritelivir ointment matching placebo
Drug: Zovirax® cream
  Arms: Zovirax® cream

SUMMARY:
Randomized, double-blind, multi-center, three arm parallel group, comparative trial to assess pritelivir ointment safety and efficacy, ie, proportion of subjects with non-ulcerative lesions, in adult subjects with recurrent herpes labialis (RHL) in comparison with placebo or Zovirax® Cream. The start of treatment with trial medication will be initiated by the subject within one hour of noticing the first sign or symptom (eg, prodrome) of a recurrence of herpes labialis. Trial medication will be applied to the affected area 5 times daily for 4 days.

After self-initiation of treatment with trial medication subjects will be assessed daily by the Investigator until complete healing for a maximum of 13 days.

Subjects will document application of trial medication and the status of their lesion in a diary. There will also be blood sampling, ECG measurement and physical examination performed at the investigational site.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women of any ethnic group aged ≥18 years ;
* Subjects should have experienced ≥4 recurrences of herpes labialis in the previous 12-months period;
* Subjects should have experienced prodromal symptoms in at least 50% of recurrent Herpes labialis (rHL) episodes and should have developed ulcerative lesions that have progressed through vesicle, ulcer, and crust stages in at least 50% of the episodes;
* Willingness not to use any topical application (such as cosmetics, lip balm, sunscreens etc…) other than the trial medication in the area of lesion development from start of prodromal symptoms to complete healing;
* Willingness not to use any systemic and topical anti-Herpes Simplex Virus (HSV) agent during the trial participation including prescription and over-the-counter (OTC) products;
* Willingness not to use any systemic, anti-inflammatory or analgesic agents from start of prodromal symptoms to healing;
* Willingness to refrain from mechanical disruption (ie, scrubbing, lancing, shaving) of the prodromal area or lesion after start of treatment with trial medication until end of the trial participation;
* Women of child bearing potential and males must use adequate contraception;
* Subject must give written informed consent.
* Subjects with current lesion may be enrolled, but they must not treat the lesion present at screening/randomization with the trial medication; they should be instructed to wait for their next subsequent lesion

Exclusion Criteria:

* Known intolerance to pritelivir or any of the ointment ingredients;
* Known intolerance to Zovirax® Cream or any of the ingredients (ie, acyclovir, cetostearyl alcohol, mineral oil, poloxamer 407, propylene glycol, sodium lauryl sulfate, and white petrolatum) or valacyclovir;
* Any skin conditions that could interfere with the assessment of herpes labialis recurrences (eg, eczema, psoriasis, acne etc…)
* Any other condition which in the opinion of the Investigator would interfere with successful completion of this clinical trial
* Pregnant and/or breastfeeding women
* Participation in any investigational drug trial within the last 30 days before randomization for this clinical trial
* Previous treatment with pritelivir tablets
* Previous participation in a HSV vaccination Trial unless having received placebo.
* Clinically relevant ECG abnormalities (eg, QTc according to Fridericia: QTcF > 450 ms for males and QTcF > 470 ms for females; PR > 220 ms) at screening.
* Clinically relevant abnormalities in laboratory indices at screening which in the opinion of the investigator might have an impact on the safety and evaluability of the subject.
* Known chronic infections which in the opinion of the investigator might have an impact on the safety and evaluability of the subject.
* Evidence of active malignancy or immunodeficiency disease, or require chronic use of immunosuppressive drugs (eg, systemic steroids) or topical steroids, or chronically use antiviral medication with activity against HSV.
* HIV positive based on screening labs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Actual)
Dates: Start 2016-11-29 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-10-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Scottsdale, Arizona
  - Santa Rosa, California
  - Pinellas Park, Florida
  - Edina, Minnesota
  - St Louis, Missouri
  - Akron, Ohio
  - Cincinnati, Ohio
  - Anderson, South Carolina
  - Greer, South Carolina
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients with labial HSV develop an outbreak only a few times per year. Therefore, more patients need to be enrolled to obtain the planned number of evaluable herpes labialis recurrences, as roughly 40% of subjects do not develop a recurrence.
  Overall, 362 subjects were enrolled and randomized. 223 started the self-initiated treatment due to an outbreak. The remaining 139 subjects did not have an outbreak and were not treated.
Groups:
- Pritelivir 5% w/w Ointment: Topical treatment (20 applications), 5 times daily for 4 days
  Pritelivir 5% w/w ointment
- Pritelivir Ointment Matching Placebo: Topical treatment (20 applications), 5 times daily for 4 days
  Pritelivir ointment matching placebo
- Zovirax® Cream: Topical treatment (20 applications), 5 times daily for 4 days
  Zovirax® cream
Period: Overall Study
Arm/Group | Pritelivir 5% w/w Ointment | Pritelivir Ointment Matching Placebo | Zovirax® Cream
Started | 73 | 73 | 77
Completed | 67 | 70 | 71
Not Completed | 6 | 3 | 6
Not completed — Lost to Follow-up | 6 | 3 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pritelivir 5% w/w Ointment | Pritelivir Ointment Matching Placebo | Zovirax® Cream | Total
Number analyzed (Participants) | 73 | 73 | 77 | 223
Age, Continuous [Median (Full Range); unit: years] | 54 [21 to 74] | 49 [20 to 77] | 51 [18 to 79] | 51 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 53 | 56 | 161
  Male | 21 | 20 | 21 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 8 | 6 | 10 | 24
  White | 63 | 65 | 65 | 193
  More than one race | 1 | 0 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 73 | 73 | 77 | 223
BMI [Median (Full Range); unit: kg/m^2] | 27.8 [19.3 to 48.5] | 27.3 [19.4 to 56.7] | 28.1 [17.1 to 47.7] | 27.8 [17.1 to 56.7]

OUTCOME MEASURES:

1. Primary Outcome: Efficacy Measured by Percentage of Subjects With Non-ulcerative Lesions Based on Principal Investigator's Assessment
Description: The Investigator assessed subjects for lesion stage at every visit as long as lesions were present from Visit 1 to the End of Trial Visit (Day 12± 1) as a maximum. Percentage of subjects with non-ulcerative lesions (i.e, scoring below 3) based on the Principal Investigators Assessment. Lesion stages were defined as follows: 1-Prodrome; 2a-Redness; 2b-Erythema-Redness; 3-Small Blister; 4-Ulcer; 5-Crust; 6-Drying up and healing; 0-Resolved
Time Frame: 13 days
Population: Primary analysis for the ITT ( intent to treat) population; multiple imputation.
Measure: Number; unit: percentage of partcipants
Arm/Group | Pritelivir 5% w/w Ointment | Pritelivir Ointment Matching Placebo | Zovirax® Cream
Number analyzed (Participants) | 71 | 72 | 75
percentage of partcipants
  Non-ulcerative recurrences | 21.8 | 16.4 | 19.9
  Ulcerative recurrences | 78.2 | 83.6 | 80.1
Statistical Analysis 1: Comparison: Pritelivir 5% w/w Ointment vs Pritelivir Ointment Matching Placebo; Test type: Superiority; p = 0.4294, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: 10 months
Description: Subjects were interviewed by the investigational site staff pre-dose and at every visit using nonleading questions.
Arm/Group | Pritelivir 5% w/w Ointment | Pritelivir Ointment Matching Placebo | Zovirax® Cream
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/73 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/73 | 0/73 | 0/77
Other Adverse Events (participants affected / at risk) | 30/73 | 27/73 | 27/77
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pritelivir 5% w/w Ointment (N=73) | Pritelivir Ointment Matching Placebo (N=73) | Zovirax® Cream (N=77)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Chapped lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Lip blister (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Application site inflammation (General disorders) | 0 (0) | 1 (1) | 0 (0)
Application site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Induration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Oral herpes (Infections and infestations) | 10 (10) | 5 (5) | 3 (3)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Limb crushing injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Blood sodium decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
C-reactive protein increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST-T change (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram T wave inversion (Investigations) | 0 (0) | 0 (0) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haptoglobin increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Urine analysis abnormal (Investigations) | 2 (2) | 0 (0) | 1 (1)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 3 (3)
Sinus headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 3 (3)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Papule (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and Investigator agree not to publish the results or other data of this Study without the prior written consent of Sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-31): https://cdn.clinicaltrials.gov/large-docs/92/NCT02871492/Prot_SAP_000.pdf